CLINICAL TRIAL: NCT00009204
Title: Serotonergic Pharmacotherapy for Agitation of Dementia
Acronym: SPAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bruce Pollock (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Bruce Pollock, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH059666-01 (NIH); R01MH059666-01 (NIH); IA0014; DSIR GT-GP; NCT00000184 (obsolete NCT alias)
Record Dates: First submitted 2001-01-23; First posted 2001-01-24 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Dementia; Alzheimer Disease; Dementia, Vascular
Keywords: Behavioral problems; Agitation
MeSH Terms: conditions — Dementia; Alzheimer Disease; Dementia, Vascular; Problem Behavior; Psychomotor Agitation | interventions — Citalopram; Perphenazine

INTERVENTIONS:
Drug: Citalopram [Celexa]
Drug: Perphenazine [Trilafon]

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, fixed dose study currently being conducted on two geropsychiatric units at Western Psychiatric Institute and Clinic. It seeks to evaluate the short-term safety and efficacy of citalopram and perphenazine in the treatment of 112 patients suffering from behavioral disturbances associated with dementia. Findings from this research may directly lead to improved acute pharmacotherapy for psychosis and behavioral problems in patients diagnosed with dementia. Improved treatment of behavioral complications with reduced side effects would reduce excess disability in patients diagnosed with dementia, allowing them to be maintained in the community for greater periods of time.

DETAILED DESCRIPTION:
The principal investigator is conducting an inpatient study at Western Psychiatric Institute and Clinic involving two medications for treatment of emotional and behavioral disturbances that may accompany dementia. In this study, 112 patients will be enrolled for up to 17 days in order to investigate the safety and effectiveness of both medications. Forty-two of these patients will be given a recently FDA-approved antidepressant medication called citalopram and 42 will receive one of our current, usual antipsychotic medications called perphenazine. An additional 28 patients will be given non-active placebo capsules. Which treatment a patient is given during the study will be determined by chance. Findings from this investigation may directly lead to the improvement of symptoms such as: agitation, hostility, suspiciousness, hallucinations, and unusual thoughts. Improved treatment of problematic behaviors and a decrease in medication-associated side effects would enable dementia patients to be cared for in their home environments for longer periods of time.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for diagnosis of dementia of the Alzheimer's type (AD), Vascular dementia (VD), mixed (AD and VD) or dementia NOS (Not Otherwise Specified)
* Presents with psychosis or behavioral problems severe enough to endanger the patient's health, well-being or safety, as evidenced by a score of at least 3 (moderate) on one of the Neurobehavioral Rating Scale (NBRS) agitation items (8,11,14) or psychosis items (16,18,20) and are not secondary to physical illness nor amenable to environmental optimization
* Able to participate in study evaluations and ingest oral medication
* Has next of kin or a guardian available to consent to patient's participation.

Exclusion Criteria:

* Has an unstable medical illness including significant cardiac (specifically bradycardia with ventricular rate below 50), renal, hepatic, or neurological illness (especially Parkinson's disease) other than dementia
* Meets DSM-IV criteria for Delirium upon admission to Western Psychiatric Institute and Clinic
* Has been medicated within 4 weeks of protocol admission with fluoxetine or 2 weeks with a monoamine oxidase inhibitor (patients will undergo a monitored psychotropic drug washout prior to entering the protocol)
* Is currently being treated with cognitive enhancing drugs (Tacrine or Aricept) or any experimental drug
* Has a concurrent diagnosis of schizophrenia, bipolar disorder, or major depression
* Has preexisting orthostatic hypotension (with > 20 mmHg change from sitting to standing pressure)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-09; Primary Completion 2000-04 (Actual); Study Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce G. Pollock, M.D., Ph.D., Principal Investigator — Western Psychiatric Institute and Clinic
Locations (1):
- University of Pittsburgh Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States